CLINICAL TRIAL: NCT04155307
Title: Is the Evaluation of Anal Distensibility by Endoflip® Technique Useful for the Diagnosis of Anismus?
Acronym: Endo-DC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018/0347/HP
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Anismus; Distal Constipation
MeSH Terms: interventions — Defecography; Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Detection of anismus in patients with distal constipation (Experimental)
  Interventions: Device: Anal EndoFLIP®; Diagnostic Test: Anal Manometry; Diagnostic Test: Defecography; Diagnostic Test: Electromyogram

INTERVENTIONS:
Device: Anal EndoFLIP® — Anal EndoFLIP® measure to evaluate anal compliance
Diagnostic Test: Anal Manometry — Anal Manometry done in standard care
Diagnostic Test: Defecography — Defecographydone in standard care
Diagnostic Test: Electromyogram — Electromyogram done in standard care

SUMMARY:
Terminal constipation affects 13 to 20% of the french population. Anismus is defined by an absence of relaxation or a paradoxical contraction of the striated anal sphincter muscle during defecation.

Anismus is one of the main causes of terminal constipation. Anismus diagnosis is retained if 2 out of 3 examinations (manometry, electromyogram, defecography) are positive.

EndoFLIP® is a new medical device developed to measure distensibility of a hollow organ. Anal EndoFLIP® l could be a more sensitive and specific tool for detecting anismus in patients with distal constipation.

60 patients suffering from distal constipation will be included in order to perform, in addition to the usual examinations, an anal EndoFlip in order to test the sensitivity and specificity of this method for the diagnosis of anismus.

ELIGIBILITY:
Inclusion Criteria:

* patient older than 18 years
* patient with distal constipation defined according to the Rome IV criteria, for at least 3 months and verified by a transit time study showing a predominant slowing of markers at the recto-sigmoid level.
* patient who read and signed the informed consent form

Exclusion Criteria:

* Patients with a predominant right of left colonic constipation;
* Pregnant woman or woman with no effective contraception and of childbearing age
* Patient with inflammatory bowel disease, ischemic colitis, history of colon or rectal cancer, infectious colitis or proctologic disease.
* Patient with anorectal malformation
* Patient with an history of pelvic floor radiotherapy
* Patient with a digestive stoma
* Insertion of the probe impossible or painful
* Patient who has participated to a clinical trial within 30 days prior to the inclusion visit
* Patient not understanding or reading French
* Patients under guardianship, curatorship, safeguard of justice
* Patient without liberty by administrative or judicial decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
Sensitivity of the anal distensibility evaluated with the EndoFLIP® technique for the diagnosis of anismus | 30 min
Specificity of the anal distensibility evaluated with the EndoFLIP® technique for the diagnosis of anismus | 30 min

CONTACTS AND LOCATIONS:
Overall Officials: Laura BRIL, MD, Principal Investigator — University Hospital, Rouen
Locations (1):
- Rouen University Hospital, Rouen, France

IPD SHARING:
Plan to Share IPD: No